CLINICAL TRIAL: NCT00334308
Title: Barley Protein and Coronary Heart Disease Risk Reduction
Brief Title: Barley Protein and CVD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REB 02-113C
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: Hypercholesterolemia; Cardiovascular Disease; Diet Therapy
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases | interventions — Caseins; Bread

INTERVENTIONS:
Procedure: Barley protein bread or control (casein) bread

SUMMARY:
The Question posed is: Does an barley protein concentrate have health benefits similar to those demonstrated for soy protein foods which would justify the use of the non-fiber components of barley as functional food ingredients? Hypotheses: 1. Cholesterol Lowering: There is good evidence indicating that soy protein lowers serum cholesterol levels. The evidence was strong enough for a health claim for coronary heart disease risk reduction to be approved by the FDA. In addition, we have found that wheat gluten significantly reduced serum triglyceride levels. However, there is a need to assess the possible health benefits other vegetable protein sources. Barley is grown in relatively large amounts in Canada and barley protein would be a readily available vegetable protein source if health attributes could be ascribed to it. In addition other components of barley, including plant sterols and phenolics, may have hypocholesterolemic and antioxidant properties. 2. Antioxidant: In addition to cholesterol-lowering and possibly of equal importance in terms of prevention of cardiovascular and other chronic diseases, the barley phenolics associated with barley protein and may have added benefits as antioxidants. 3. Markers of Inflammation: Barley components are considered to be hypoallergenic. Hence their use in the cosmetic industry. Auto-immune and inflammatory responses are associated with increased CHD risk. Barley protein consumption may therefore reduce the levels of the pro-inflammatory cytokines; and the acute phase proteins. 4. Arterial Dilatation: Barley proteins may also have beneficial effects on vascular reactivity which may reduce CHD risk on account of their higher arginine:lysine ratio. Arginine enhances nitric oxide synthesis associated with endothelial relaxation and arterial dilatation. Barley may therefore increase pulmonary nitric oxide levels.

DETAILED DESCRIPTION:
Design: The effect of oat protein extract will be assessed in one-month feeding studies of forty healthy men and women with raised serum cholesterol levels. Two breads will be prepared, one control and one providing 45 g/d barley protein to be fed for one month each in a randomized crossover design.

Diets: The diets will be the subjects' usual diets which appropriately will be NCEP Step 2 diets for patients treated without medications with this degree of hyperlipidemia. Those who are not on an NCEP Step 2 diet will be instructed accordingly. During the first phase, the two one-week recorded diets for each patient will be photocopied and returned to the patient to be used as the dietary model for the subsequent period. We have found that this approach is effective in stabilizing the diets in our soy protein studies. Supplements: Will be breads with test and control supplements providing the identical daily energy intake. The increase in protein in the barley supplements will be matched by the use of protein from milk protein (casein). Similarly the increased polyunsaturated, monounsaturated and saturated fatty acids in the test supplement will be matched by addition of an appropriate blend of oils in the control. Baked goods will be prepared at our clinic and a seven-day supply will be provided to each participant at the beginning of each week. The exact formulation of the supplements will involve product development, palatability testing and chemical analysis of the prototypes in the initial phase of the study. Compliance: compliance will be assessed from completed weekly diet records where supplement intake is recorded daily. These records will be reviewed by a dietitian with the subject at the end of the week. In addition, uneaten supplements will be returned, weighed and noted on the menu plans by the dietitian. Diet records will also be assessed to ensure the predetermined diet plan is followed according to the phase one recorded diet.

ELIGIBILITY:
Inclusion Criteria:

* men and postmenopausal women with mild- to-moderate hypercholesterolemia
* Body mass index >18 kg/m2 and < 36 kg/m2.
* treated by diet
* Alcohol intake < 14 drinks per week.
* Fasting plasma triglyceride (TG) concentration > 0.5 mmol/l and < 4.5 mmol/l.
* Fasting plasma LDL cholesterol concentration > 3.5 mmol/l at diagnosis.

Exclusion Criteria:

* Child-bearing women
* Taking cholesterol lowering medications at the start of the study, unless their LDL-cholesterol levels are >3.5 mmol/L.However, with their physician's approval those who wish to join but are already taking cholesterol lowering medications with low LDL-cholesterol levels (e.g. <2.5 mmol/L) may join the study providing the medications are stopped for one month.
* Change the type or dose of their drug treatment during the study
* Patients judged as having a likelihood of being non-compliant with instructions for whatever reason
* Food allergies
* Evidence or history of diabetes, renal liver disease or gastrointestinal disease
* Recent (within 6 months)) major cardiovascular event (stroke or myocardial infarction)
* Secondary causes of hypercholesterolemia (or untreated hypothyroidism)
* Uncontrolled blood pressure
* Major disability or disorder such as liver disease, renal failure or cancer or with major surgery < 6 months prior to randomization

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)

PRIMARY OUTCOMES:
total and LDL cholesterol, LDL:HDL cholesterol ratio

SECONDARY OUTCOMES:
Blood pressure, HDL cholesterol, HDL2 and HDL3, triglyceride, apolipoprotein A1 and B, Lp(a) and LDL particle size; oxidative stress,inflammatory biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: David JA Jenkins, MD, Principal Investigator — University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jenkins DJ, Srichaikul K, Wong JM, Kendall CW, Bashyam B, Vidgen E, Lamarche B, Rao AV, Jones PJ, Josse RG, Jackson CJ, Ng V, Leong T, Leiter LA. Supplemental barley protein and casein similarly affect serum lipids in hypercholesterolemic women and men. J Nutr. 2010 Sep;140(9):1633-7. doi: 10.3945/jn.110.123224. Epub 2010 Jul 28. PMID 20668250